CLINICAL TRIAL: NCT02985320
Title: A Open-label Phase I Study to Evaluate Safety of a Sabin Inactivated Poliovirus Vaccine (sIPV) in Adults, Children, and Infants, and a Blinded, Randomized and Controlled Phase II to Evaluate Safety and Immunogenicity of it in Infants
Brief Title: Studies of the Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-sIPV-1001
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Poliomyelitis
Keywords: Sabin strain; Inactivated poliovirus vaccine; poliomyelitis; safety; immunogenicity; infant
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- Phase I Adult Group - High dosage (Experimental): * Single intramuscular injection of the investigational vaccine(0.5 ml) on Day 0;
  * Intervention: Single-dose regimen of high dosage investigational sIPV
  Interventions: Biological: Single-dose regimen of high dosage investigational sIPV
- Phase I Adult Group - Medium dosage (Experimental): * Single intramuscular injection of the investigational vaccine(0.5 ml) on Day 0;
  * Intervention: Single-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: Single-dose regimen of medium dosage investigational sIPV
- Phase I Child Group - High dosage (Experimental): * Single intramuscular injection of the investigational vaccine(0.5 ml) on Day 0;
  * Intervention: Single-dose regimen of high dosage investigational sIPV
  Interventions: Biological: Single-dose regimen of high dosage investigational sIPV
- Phase I Child Group - Medium dosage (Experimental): * Single intramuscular injection of the investigational vaccine(0.5 ml) on Day 0;
  * Intervention: Single-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: Single-dose regimen of medium dosage investigational sIPV
- Phase I Infant Group - High dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of high dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of high dosage investigational sIPV
- Phase I Infant Group - Medium dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of medium dosage investigational sIPV
- Phase I Infant Group - Low dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of low dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of low dosage investigational sIPV
- PhaseⅡExperimental Group - High dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of high dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of high dosage investigational sIPV
- PhaseⅡExperimental Group - Medium dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of medium dosage investigational sIPV
- PhaseⅡExperimental Group - Low dosage (Experimental): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of low dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of low dosage investigational sIPV
- PhaseⅡControl Group -commercialized sIPV (Active Comparator): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention:Three-dose regimen of commercialized sIPV
  Interventions: Biological: Three-dose regimen of commercialized sIPV
- PhaseⅡ Control Group -commercialized IPV (Active Comparator): * Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively;
  * Intervention: Three-dose regimen of commercialized IPV
  Interventions: Biological: Three-dose regimen of commercialized IPV

INTERVENTIONS:
Biological: Single-dose regimen of high dosage investigational sIPV — The investigational vaccines were manufactured by Sinovac Biotech Co., Ltd..
  Arms: Phase I Adult Group - High dosage; Phase I Child Group - High dosage
Biological: Single-dose regimen of medium dosage investigational sIPV — The investigational vaccines were manufactured by Sinovac Biotech Co., Ltd..
  Arms: Phase I Adult Group - Medium dosage; Phase I Child Group - Medium dosage
Biological: Three-dose regimen of high dosage investigational sIPV — The investigational vaccines were manufactured by Sinovac Biotech Co., Ltd..
  Arms: Phase I Infant Group - High dosage; PhaseⅡExperimental Group - High dosage
Biological: Three-dose regimen of medium dosage investigational sIPV — The investigational vaccines were manufactured by Sinovac Biotech Co., Ltd..
  Arms: Phase I Infant Group - Medium dosage; PhaseⅡExperimental Group - Medium dosage
Biological: Three-dose regimen of low dosage investigational sIPV — The investigational vaccines were manufactured by Sinovac Biotech Co., Ltd..
  Arms: Phase I Infant Group - Low dosage; PhaseⅡExperimental Group - Low dosage
Biological: Three-dose regimen of commercialized sIPV — The control vaccine was manufactured by Chinese Academy of Medical Sciences.
  Arms: PhaseⅡControl Group -commercialized sIPV
Biological: Three-dose regimen of commercialized IPV — The control vaccine was manufactured by Sanofi Pasteur S.A (IMOVAX POLIO).
  Arms: PhaseⅡ Control Group -commercialized IPV

SUMMARY:
The purpose of this study is to evaluate the safety of sIPVs of different dosages in adults, children and infants in a phase I open-label study, and then assess its immunogenicity and safety in healthy infants between 60 and 90 days old in a phase II blind, randomized, and controlled study.

DETAILED DESCRIPTION:
This study is a combination of phases I and II. Phase I study is open-label, and only collect safety information of the investigational sIPVs in adults, children and infants. Phase II study is double-blind, randomized, controlled study of the immunogenicity and safety of the investigational vaccines and two other commercialized inactivated poliovirus vaccines in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 60-90 days old, 6-12 years old, or 18-49 years old;
* Healthy volunteers who fulfill all the required conditions for receiving the investigational vaccine as established by medical history and clinical examination and determined by investigators;
* Proven legal identity;
* Participants (≥ 18 years old), or guardians of the participants (< 18 years old) should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;
* Axillary temperature ≤ 37.0 °C;

Exclusion Criteria:

* Breast feeding, pregnant, or expected to conceive in the next 60 days;
* History of allergy to any vaccine, or any ingredient of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* serious chronic diseases, serious cardiovascular disease, hypertension or diabetes that cannot be stabilized by medication, liver or kidney disease, malignancy, etc;
* severe nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* History of thyroidectomy, asplenia, functional asplenia, or any condition resulting in the absence or removal the spleen;
* Bleeding disorder diagnosed by a doctor (e.g., coagulation factor deficiency, coagulation disorder, or platelet disorder) , or significant bruising or coagulopathy;
* Long term history of alcoholism or drug abuse;
* Receipt of any of the following products:

  1. Any subunit or inactivated vaccine within the past 7 day;
  2. Any live attenuated vaccine within the past 14 days;
  3. Any other investigational medicine(s) within the past 30 days;
  4. Any blood product within the past 3 months;
  5. Any immunosuppressant, cytotoxic medications, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within the past 6 month prior to study entry;
* Acute illness or acute exacerbation of chronic disease within the past 7 days;
* Axillary temperature > 37.0 °C;
* Infant participants with prior vaccination of poliovirus;
* Any other factor that, in the judgment of the investigator, suggesting the volunteer is unsuitable for this study;

Ages: 2 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 708 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of each group of the phase II trial after three-dose regimen | 90 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.
The post-immune geometric mean titer (GMT) of each group of the phase II trial after three-dose regimen | 90 days
  GMT of each group of the phase II trial 30 days after three-dose regimen which lasts 60 days.
The geometric mean fold increase (GMI) of each group after three-dose regimen | 90 days
  The GMI is the increase of post-immune GMT from pre-immune GMT.

SECONDARY OUTCOMES:
The incidences of solicited adverse events (AEs) of each group in both phase I and II trials | 7 days
  Solicited AEs occurred within 7 days after each injection will be collected.
The incidences of unsolicited adverse events (AEs) of each group in both phase I and II trials | 30 days
  Unsolicited AEs occurred within 30 days after each injection will be collected.
The incidences of serious adverse events (SAEs) of each group in both phase I and II trials | 30 days
  SAEs occurred within 30 days after each injection will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Pizhou City Center for Disease Control and Prevention, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu K, Ying Z, Wang L, Hu Y, Xia J, Chen L, Wang J, Li C, Zhang Q, Gao Q, Hu Y. Safety and immunogenicity of inactivated poliovirus vaccine made from Sabin strains: A phase II, randomized, dose-finding trial. Vaccine. 2018 Oct 29;36(45):6782-6789. doi: 10.1016/j.vaccine.2018.09.023. Epub 2018 Sep 21. PMID 30249424